CLINICAL TRIAL: NCT04519060
Title: An Eye-opener: The Impact of Eye Shields for Infants After Dilated Exam
Brief Title: Eye Shields for Infants After Dilated Exam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Maxine Ogbaa, BSN, Children's Hospital Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-20-00211
Record Dates: First submitted 2020-05-17; First posted 2020-08-19 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Infant, Newborn, Disease; Pain; Retinopathy of Prematurity; Eye Diseases
Keywords: eye shield; eye protector; eye patch; eye mask; phototherapy
MeSH Terms: conditions — Disease; Pain; Retinopathy of Prematurity; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No eye shields after dilated eye exam (No Intervention): Eye dilation for scheduled exam will be followed by routine clinical care.
- Eye shields after dilated eye exam (Experimental): Eye dilation for scheduled exam will be followed by routine clinical care and the application of eye shields. They will be worn until four (4) hours after the last dose of dilating eye drops.
  Interventions: Device: phototherapy eye shield

INTERVENTIONS:
Device: phototherapy eye shield — Phototherapy eye shields will be applied to the eyes of infants dilated for scheduled eye exam. They will be worn until four (4) hours after the last dose of dilating eye drops.
  Other Names: phototherapy eye protector; phototherapy eye mask
  Arms: Eye shields after dilated eye exam

SUMMARY:
The eyes of hospitalized infants are often assessed by dilated exam, and there is evidence that infants experience post-exam stress. Investigators will evaluate whether eye shields for infants after dilated eye exam lessen stress and discomfort.

DETAILED DESCRIPTION:
Neonatal eye examinations are the standard of best practice in pediatrics. In the acute clinical setting, infants' eyes are inspected for eye development, defect, and disease. There is anecdotal and clinical evidence that infants experience stress after eye dilation. Investigators will evaluate whether eye shields for infants after dilated eye exam lessen stress and discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Chronological age 0-12 months
* Infants who require dilated eye exams
* Parent or legal guardian consent/permission granted

Exclusion Criteria:

* More than a two-week interval between dilated eye exams
* Prior or ongoing medical treatment or therapy for the eye(s)
* Functional blindness diagnosed by eye exam

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of stress events | 4-6 hours (from first dose of eye dilating medication to four hours after last dose)
  The primary outcome will be measured by the count of apneas and bradycardias (stress events) experienced by the infant during the period of eye dilation without eye shields as compared to the total stress events experienced when dilated eyes are covered with eye shields.

SECONDARY OUTCOMES:
Number of stress events amongst covariates | 4-6 hours (from first dose of eye dilating medication to four hours after last dose)
  The secondary outcome measure will be abstracted from covariate data (e.g., infant gestational age at birth, post-natal age, weight, and ventilation status) to assess the influence of covariables on the response to eye shields as an intervention to lessen stress and discomfort in hospitalized infants after dilated eye exam.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No